CLINICAL TRIAL: NCT02269891
Title: A Randomized Double-Blind, Placebo-Controlled, Parallel Clinical Trial on the Efficacy of a Combination Herbal Product, Biotropics' Nu Femme, on Menopausal Symptoms and Quality of Life in Women
Brief Title: A Clinical Trial on the Efficacy of a Combination Herbal Product, Biotropics' Nu Femme, on Menopausal Symptoms and Quality of Life in Women
Acronym: 14NMHB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Biotropics Malaysia Berhad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14NMHB
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Menopausal Symptoms
Keywords: Menopausal symptoms; Peri-menopause; Nu Femme; Labisia pumila; Eurycoma longifolia; Hot flash; Joint pain
MeSH Terms: conditions — Hot Flashes; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Nu Femme (Experimental): Two capsules (500mg total) taken once daily in the morning after breakfast for 24 weeks
  Interventions: Dietary Supplement: Nu Femme
- Placebo (Placebo Comparator): Two capsules taken once daily in the morning after breakfast for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nu Femme — Combination product of Labisia pumila and Eurycoma longifolia extracts
  Arms: Nu Femme
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of an herbal combination product called Nu Femme, on menopausal symptoms in peri-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Female of any race between the ages of 40 and 55 years (inclusive)
* Experiencing perimenopause (irregular menstrual cycles (>3 months) or cessation of menstrual period for at least 3 months within the last 12 months) OR women in menopause (cessation of menstrual period for at least 12 months).
* Peri-menopausal women must have an endometrial stripe < 8 mm by ultrasound at screening and menopausal women must have an endometrial stripe < 5 mm. Not required for subjects without an intact uterus.
* Women with an intact cervix must have a pap smear that is normal within 12 months of screening.
* Experiences menopausal transition symptoms such as hot flushes, sweating, sleep disturbance, migraine, anxiety, vaginal dryness and sexual problems.
* Minimum of 4 hot flashes per day or 28 per week
* Total scores of Menopause Rating Scale ≥17 indicating the menopausal symptoms are moderate or severe
* TSH screening to exclude undiagnosed hyperthyroidism
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements.

Exclusion Criteria:

* Women with a positive mammogram
* Significant cardiac history including uncontrolled hypertension (defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg) or current diagnosis of any major diseases of the cardiovascular, hepatic, renal, gastrointestinal, pulmonary or endocrine systems
* Uncontrolled hyperlipidemia
* History or current diagnosis of breast cancer or breast cancer in an identical twin, or any cancer (except non-melanomatous skin cancer) diagnosed less than 5 years prior to randomization. Subjects with other cancers in full remission more than 5 years after diagnosis are acceptable with the exceptions of breast cancer or genital organ cancer (e.g., cervical cancer, uterine cancer, endometrial cancer, or ovarian cancer)
* Uncontrolled diabetes (Type I or Type II)
* Uncontrolled and/or untreated thyroid disorder
* History or current diagnosis of any major diseases of the cardiovascular, hepatic, renal, gastrointestinal, pulmonary or endocrine systems
* History or current diagnosis of autoimmune conditions, immunodeficiency or gynaecological disease
* Clinically significant mental depression that is not well-controlled in the opinion of the investigator
* Subject has undergone major surgery within the past one year prior to the randomization visit, except cholecystectomy, and appendectomy
* Subject smokes more than 15 cigarettes a day
* History of alcohol or drug abuse within the past year
* Subject has demonstrated non-compliance with treatment while enrolled in other experimental protocols to which the Investigator has knowledge
* Subject has a mental disability or significant mental illness, legal incapacity or limited legal capacity or any other lack of fitness, in the Investigator's opinion, to preclude subject's participation in or to complete the study
* History or findings of undiagnosed abnormal vaginal bleeding within the previous two years prior to the randomization visit, including conditions that, in the Investigator's opinion are likely to be the source of unpredictable vaginal bleeding (i.e. leiomyoma or endometrial polyps)
* Subject has uterine fibroids (> 2cm) or endometriosis. This assessment will be based on the size of the uterus of each participant and will be assessed by the Qualified Investigator
* Pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Positive urine pregnancy test result
* Polycystic ovary syndrome (PCOS)
* History of abnormal Pap smear
* Significant abnormal liver function as defined as AST and/or ALT > 2 x the upper limit of normal (ULN), and/or bilirubin > 2 x the ULN
* eGFR <60
* Bleeding disorders or anaemia of any etiology defined as haemoglobin ≤ 110 g/L
* Subject has taken any of the following medications in the time periods specified prior to the screening visit and during the study

Sex hormones:

Vaginal rings and vaginal creams, ointments or gels 1 week Transdermal or topical 4 weeks DHEA within 24 weeks Natural supplements advertised to have hormonal effects within 4 weeks Oral within 4 weeks Intrauterine progestin implants within 8 weeks Progestin implants and estrogen alone injections within 12 weeks Injected progestin and estrogen or androgen implants or pellets within 24 weeks

Gonadotropin-releasing hormone (GnRH) agonists within 24 weeks

Selective Estrogen Receptor Modulators (SERMs) within 4 weeks

Glucocorticoids - Chronic high dose (≥ 7.5 mg prednisone per day or equivalent) for the past 12 weeks. Exceptions: Chronic low dose corticosteroid use (< 7.5 mg prednisone per day, or equivalent) is permitted provided the subject has been stabilized on a dose for at least 12 weeks prior to randomization and maintains the current dose and dosing regimen during the study. Acute topical, inhaled, or oral (e.g. dose packs) use is not exclusionary and will be permitted during the course of the study.

Antidepressant and/or antianxiety medications within 4 weeks unless a chronic stable dose has been maintained for greater than 12 weeks. Subject must maintain current dose and dosing regimen during the study. Use of Effexor (Venlafaxine HCl) within 4 weeks is exclusionary. Use of Dixarit (Clonidine HCl) within 2 weeks is exclusionary.

Thyroid or anti-epileptic medications within 12 weeks unless a chronic stable dose has been maintained for greater than 12 weeks prior to randomization. Subjects must maintain current dose and dosing regimen during the study

Use of Prostaglandins within 4 weeks

Other investigational study medications within 4 weeks

Current use of propranolol

Current use of an intrauterine device (IUD)

Use of natural health products, such as primrose oil, black cohosh, soy products, other than vitamin and/or mineral supplements within 4 weeks

* Known allergy or hypersensitivity to study product ingredients
* Subjects on a weight reduction program or a medically supervised diet.
* Unexplained weight loss or weight gain of more than 5 kg in the month prior to randomization
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2014-10; Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of hot flashes | Baseline to week 12
  Assessed based on hot flash symptoms score

SECONDARY OUTCOMES:
Frequency and severity of joint pain | Baseline to week 12
  Assessed based on joint pain symptoms score
Frequency and severity of hot flashes | Baseline to week 24
  Assessed based on hot flash symptoms score
Frequency and severity of hot flashes | Week 12 to week 24
  Assessed based on hot flash symptoms score
Frequency and severity of joint pain | Baseline to week 24
  Assessed based on joint pain symptoms score
Frequency and severity of joint pain | Week 12 to week 24
  Assessed based on joint pain symptoms score
Health related quality of life | Baseline to weeks 3, 6, 12 and 24
  Assessed using the Menopause Rating Scale (MRS)
Menopause specific quality of life | Baseline to weeks 3, 6, 12 and 24
  Assessed using the Menopause Specific Quality of Life questionnaire (MENQOL)
Serum hormone concentrations | Baseline to week 12
  Estradiol-17b, FSH, LH, total testosterone and free testosterone
Serum Lipid Profile | Baseline to week 12
  Total cholesterol, HDL-C, LDL-C and triglycerides

OTHER OUTCOMES:
Bone markers | Baseline to week 12
  NTX and BSALP
Blood safety parameters | Baseline to week 12
  CBC, electrolytes (Na K CL), glucose, creatinine, BUN, AST, ALT, GGT, bilirubin, Ca, albumin
Pap smear | Baseline to week 12
  Histological analysis for abnormal cells
Pelvic ultrasound | Baseline to week 12
  To determine changes in endometrial thickness
Incidence of adverse events | Baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (4):
- Canada (4):
  - KGK Synergize Inc., London, Ontario
  - Manna Research - Toronto, Toronto, Ontario
  - Manna Research - Quebec, Lévis, Quebec
  - Manna Research - Montreal, Pointe-Claire, Quebec